CLINICAL TRIAL: NCT04096820
Title: Protocol 19-01: Canadian, Single Centre, Pilot, Open Label Study to Evaluate the Efficacy and Safety of the Bacterial Vaccine Uromune in Treating Recurrent Urinary Tract Infections in Women.
Brief Title: Uromune in Treating Recurrent Urinary Tract Infections in Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Convenience sample based on available funding. Increased Covid-related costs of clinical research resulted in early termination
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. J. Curtis Nickel, Professor or Urology, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6026618
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Uti
MeSH Terms: conditions — Urinary Tract Infections | interventions — uromune

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): Uromune will be taken by the participant for 90 days.
  Interventions: Biological: Uromune

INTERVENTIONS:
Biological: Uromune — 2 sprays of vaccine under the tongue for 90 days. Liquid is to held under tongue for 2 minutes without swallowing.

SUMMARY:
To determine the effectiveness and safety of the vaccine Uromune in Canadian women with recurrent urinary tract infection.

DETAILED DESCRIPTION:
The proposal is for a real life clinical practice study in which female participants with a predefined history of recurrent UTIs in the previous year will be treated with 3 months of oral vaccine with a further 9 months of follow-up. The primary outcome will be no UTI in the 9 month efficacy period following completion of the vaccine (definition of a responder). A clinically significant and important outcome will be defined as a responder rate of 50% (50% of participants who had at least 3 UTIs in the previous year reporting no UTIs after therapy initiated.

ELIGIBILITY:
Inclusion Criteria:

* Can provide written consent and willingness to comply with all aspects of study treatment and study requirements.
* Individuals who have had at least 3 episodes of a UTI in the past 12 months or 2 UTI episodes in the past 6 months. At least one of the UTI episodes must be associated with a positive urine culture with a traditional uropathogen including Escherichia coli, Proteus spp. Staphyloccous sp. Enterococcus sp. Klebsiella sp. or Pseudomonas aeruginosa.
* Post-menopausal for a minimum of 1 year or negative pregnancy test if participant is of child bearing potential and agreement to acceptable contraceptive use from Screening Visit 1 to final follow up visit if participant is sexually active. Medically acceptable methods of contraception include hormonal contraception (i.e. estrogen, and/or progesterone or preparations that contain a combination of these hormones), non-hormonal intrauterine device or double barrier method (i.e. condom with foam or vaginal spermicidal suppository, or diaphragm with spermicide) or vasectomy of sole sexual partner. Complete abstinence alone can be used as a method of contraception.
* Free of a urinary tract infection at the time of trial inclusion.

Exclusion Criteria:

* History of bladder tumours including uterine, cervical, vaginal or urethral cancer.
* Worrisome post-voiding residual (investigator's discretion).
* Infection related to urinary lithiasis.
* Any immunological disease requiring active therapy.
* Currently receiving Immunotherapy.
* Taking any prophylactic antibiotics at screening. Any prophylactic antibiotics must be stopped the day of the screening visit.
* Any known intolerance to the ingredients of the Uromune® Immunotherapy.
* Have any other condition or disease which, in the opinion of the investigator, could compromise participant safety or interfere with the participant's participation in the study or in the evaluation of the study results.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Curtis Nickel, MD, FRCS, Principal Investigator — Professor of Urology
Locations (1):
- Centre for Advanced Urological Research, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 67 (67 subjects signed consent)
Completed | 64 (65 participants in safety group 64 participants analyzed in modified intention to treat)
Not Completed | 3
Not completed — Did not return for intervention | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated because of Covid related delay and problems with enrollment as well as cost considerations (funds ran out).
Arm/Group | Open Label
Number analyzed (Participants) | 64
Age, Continuous [Mean (Full Range); unit: years] — Eligible Age - Amendment to allow maximum age of participants to be 80 years.
  years | 56 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 64

OUTCOME MEASURES:

1. Primary Outcome: Complete Responder
Description: Participant considered complete responder if no UTI requiring antibiotics reported in the 9 month efficacy period following completion of 3 month vaccine therapy.
Time Frame: 12 months
Population: intention to treat participants received at least one dose of vaccine and had first 3-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 64
Participants | 26

2. Secondary Outcome: Number of UTI in the Efficacy Period
Description: The number of UTI in individual participants requiring antibiotics in the 9 month efficacy period following completion of vaccine therapy will be compared to the number of UTIs requiring antibiotics before therapy is initiated.
Time Frame: 12 months
Population: Modified intention to treat included all participants who received at least one dose of vaccine and had first 3-month follow-up visit
Measure: Mean (Full Range); unit: Number of UTI/month
Arm/Group | Open Label
Number analyzed (Participants) | 64
Number of UTI/month | 0.14 [0 to 20]

ADVERSE EVENTS:
Time Frame: 15 months
Description: One patient died (unrelated myocardial infarction) before the first assessment so was not included in the modified intention to treat analysis.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 1/65
Serious Adverse Events (participants affected / at risk) | 13/65
Other Adverse Events (participants affected / at risk) | 9/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=65)
Pregancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Not related to intervention
Mastectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Not related to study intervention
Colitis (Gastrointestinal disorders) | 1 (1) — Not related to study intervention
Throidectomy (Endocrine disorders) | 1 (1) — Not related to study intervention
Knee replacement (Surgical and medical procedures) | 1 (1) — Not related to study intervention
Upper GI bleed (Gastrointestinal disorders) | 1 (1) — Not related to study intervention
rectal prolapse (Gastrointestinal disorders) | 1 (1) — Not related to study intervention
hip fracture (Injury, poisoning and procedural complications) | 1 (1) — Not related to study intervention
radial bone fracture (Injury, poisoning and procedural complications) | 1 (1) — Not related to study intervention
Accidental overdose of pain medication (Injury, poisoning and procedural complications) | 1 (1) — Not related to study intervention
rib fracture (Injury, poisoning and procedural complications) | 1 (1) — Not related to study intervention
antibiotic related anaphylaxis (Immune system disorders) | 1 (1) — Not related to study intervention
Myocardial infarction (Cardiac disorders) | 1 (1) — Not related to study intervention. Result was mortality. Not unexpected.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=65)
Gastrointestinal events (Gastrointestinal disorders) | 4 (4) — GI reflux, upper GI discomfort (X2), lower abdominal burning discomfort,
rash (Skin and subcutaneous tissue disorders) | 6 (9) — mild burning of lips, burning eyes, rash left eye, rash left elbow, tingling perineum, sensitive teeth, rash left hand, burning sensation tongue, itchiness forearm
fatigue (General disorders) | 1 (1) — fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT04096820/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04096820/ICF_001.pdf